CLINICAL TRIAL: NCT02930005
Title: A Pilot Open-label Trial of Pentosan Polysulfate Sodium and Meclofenamic Acid As Adjunctive Treatments in Patients With Psychotic Disorders
Brief Title: Pentosan Polysulfate Sodium and Meclofenamic Acid as Treatments in Patients With Psychotic Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-15-0329
Record Dates: First submitted 2016-09-28; First posted 2016-10-11 (Estimated); Results first posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2018-02

CONDITIONS: Psychotic Disorders; Schizophrenia; Schizoaffective Disorder; Bipolar Disorder
Keywords: Psychotic; Schizophrenia; Schizoaffective; Bipolar
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Bipolar Disorder; Mental Disorders | interventions — Meclofenamic Acid; Pentosan Sulfuric Polyester

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Meclofenamic acid (Experimental): 150mg meclofenamic acid daily for 8 weeks
  Interventions: Drug: Meclofenamic acid
- Pentosan polysulfate sodium (Experimental): 300mg of pentosan polysulfate sodium daily for 8 weeks
  Interventions: Drug: Pentosan polysulfate sodium

INTERVENTIONS:
Drug: Meclofenamic acid
  Other Names: Meclomen
  Arms: Meclofenamic acid
Drug: Pentosan polysulfate sodium
  Other Names: Elmiron; Hemoclar; Fibrase; Anarthron
  Arms: Pentosan polysulfate sodium

SUMMARY:
This study evaluates the feasibility of administering meclofenamic acid or pentosan polysulfate sodium as an adjunctive treatment to patients diagnosed with a psychotic disorder. Half of participants will receive meclofenamic acid, while the other half will receive polysulfate sodium.

DETAILED DESCRIPTION:
Chronic, low-grade brain inflammation is involved in the development of schizophrenia and other psychotic disorders. Medications with anti-inflammatory properties, like meclofenamic acid and pentosan polysulfate may help to reduce brain inflammation and serve as a treatment of psychotic disorders.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia, schizoaffective disorder, schizophreniform disorder, bipolar I disorder, delusional disorder, other specified schizophrenia spectrum and other psychotic disorders, unspecified schizophrenia spectrum and other psychotic disorders
* Negative pregnancy test in females of childbearing age

Exclusion Criteria:

* Urine drug screen positive for psychostimulants such as cocaine, amphetamines and ecstasy
* Any infection, neoplasm, autoimmune disease or other primary inflammatory condition (3) Previous diagnosis of intellectual disability or dementia
* Current treatment with heparin
* Use of or allergy to non-steroidal anti-inflammatory agent or pentosan polysulfate sodium
* Current or anticipated corticosteroid use
* History of peptic ulcer disease, gastro esophageal reflux disease, or gastrointestinal bleeding
* Those on warfarin or any anticoagulant
* Current treatment with lithium or asthma medication
* Individuals with pre-existing liver, cardiac, or kidney disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2015-08-07; Primary Completion 2016-10-06 (Actual); Study Completion 2016-10-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Meclofenamic Acid: 150mg meclofenamic acid daily for 8 weeks
  Meclofenamic acid
- Pentosan Polysulfate Sodium: 300mg of pentosan polysulfate sodium daily for 8 weeks
  Pentosan polysulfate sodium
Period: Overall Study
Arm/Group | Meclofenamic Acid | Pentosan Polysulfate Sodium
Started | 2 | 6
Completed 2 Weeks | 2 | 2
Completed (Completed the 8 week study) | 1 | 1
Not Completed | 1 | 5
Not completed — Lost to Follow-up | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Meclofenamic Acid | Pentosan Polysulfate Sodium | Total
Number analyzed (Participants) | 2 | 6 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 6 | 8
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.5 (3.5) | 26 (8.6) | 24.6 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 2 | 4 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 6 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Cognitive Function as Assessed by the NIH Toolbox Cognitive Test Battery (NCTB) Composite Score
Description: A higher composite score on the NCTB indicates better cognitive performance. The NCTB consists of 7 tests and 8 sub-scores, and the NIH Toolbox software calculates total composite score by averaging the normalized scores of each subscale and then deriving scale scores. The "NIH Toolbox Scoring and Interpretation Guide" (found online) doesn't indicate a total composite score range (because the score ranges are infinite), but describes scoring as follows: To get a normalized composite score, the score of the test taker is compared to the scores in the NIH Toolbox nationally representative normative sample. The mean score is 100 and the standard deviation (SD) is 15. A score at or near 100 indicates average ability compared with others. Scores around 115 suggest above-average ability. Scores around 130 suggest superior ability (in the top 2 percent nationally). A score around 85 suggests below-average ability. A score in the range of 70 or below suggests significant impairment.
Time Frame: baseline, 8 weeks
Measure: Number; unit: score
Arm/Group | Meclofenamic Acid | Pentosan Polysulfate Sodium
Number analyzed (Participants) | 1 | 1
score | 31.96 | 0.96

2. Secondary Outcome: Change in Severity of Psychotic Symptoms as Assessed by Positive and Negative Syndrome Scale (PANSS)
Description: Change in the Positive and Negative Syndrome Scale (PANSS) total score after 8 weeks. The range of scores on the PANSS is 30 to 210, with higher scores associated with better outcomes.
Time Frame: baseline, 8 weeks
Measure: Number; unit: score
Arm/Group | Meclofenamic Acid | Pentosan Polysulfate Sodium
Number analyzed (Participants) | 1 | 1
score | -11 | -22

ADVERSE EVENTS:
Time Frame: up to 8 weeks
Arm/Group | Meclofenamic Acid | Pentosan Polysulfate Sodium
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/6
Other Adverse Events (participants affected / at risk) | 0/2 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Meclofenamic Acid (N=2) | Pentosan Polysulfate Sodium (N=6)
Hyperglycemia (Endocrine disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes